CLINICAL TRIAL: NCT04879121
Title: A Phase II Basket Study of the Oral TRK Inhibitor Larotrectinib (BAY2757556) in Subjects With NTRK Amplification Positive and Pan-TRK Positive Tumors
Brief Title: Larotrectinib for the Treatment of NTRK Amplification Positive, Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0564; NCI-2021-00338 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0564 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-01; First posted 2021-05-10 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Locally Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — larotrectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (larotrectinib sulfate) (Experimental): Patients receive larotrectinib sulfate PO BID on days 1-28. Cycles repeat every 28 days in the absence of unacceptable toxicity. Patients who experience disease progression and are deriving clinical benefit from larotrectinib may continue treatment per physician discretion.
  Interventions: Drug: Larotrectinib Sulfate

INTERVENTIONS:
Drug: Larotrectinib Sulfate — Given PO
  Other Names: ARRY 470 Sulfate; LOXO 101 Sulfate; LOXO-101 Sulfate; Vitrakvi

SUMMARY:
This phase II trial studies the effect of larotrectinib in treating patients with NTRK gene amplification positive solid tumors that have spread to nearby tissues or lymph nodes (locally advanced) or other places in the body (metastatic). Larotrectinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine overall response rate (ORR) to larotrectinib sulfate (larotrectinib) in patients with advanced solid tumors harboring NTRK amplification and pan-TRK expression by immunohistochemistry (IHC), calculated as the proportion of subjects with confirmed complete (CR) or partial response (PR) as best response and as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 and Response Assessment in Neuro-Oncology (RANO) criteria in primary central nervous system (CNS) tumor.

SECONDARY OBJECTIVES:

I. To evaluate the duration of response (DOR) in subjects with CR or PR as best response.

II. To estimate the proportion of subjects with any tumor regression as best response.

III. To evaluate the growth modulation index (GMI) following initiation of larotrectinib.

IV. To evaluate overall (OS) and progression-free survival (PFS) following initiation of larotrectinib.

V. To evaluate the clinical benefit rate (CBR) based on the proportion of subjects with best response of CR, PR, or stable disease lasting >= 16 weeks following initiation of larotrectinib safety.

VI. To assess the safety profile and tolerability of larotrectinib.

EXPLORATORY OBJECTIVES:

I. To characterize NTRK1, NTRK2, and NTRK3 amplification by next-generation sequencing of tumor biopsies.

II. To characterize TRKA, TRKB, and TRKC signaling in fresh pre-treatment tumor biopsies, with the aim of elucidating TRK biology and modifiers of response to larotrectinib.

III. To characterize concurrently activated oncogenic pathways in fresh pre-treatment tumor biopsies, with the aim of elucidating TRK biology and modifiers of response to larotrectinib.

OUTLINE:

Patients receive larotrectinib sulfate orally (PO) twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of unacceptable toxicity. Patients who experience disease progression and are deriving clinical benefit from larotrectinib may continue treatment per physician discretion.

After completion of study treatment, patients are followed up at 4 weeks, and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* At least 16 years of age
* Locally-advanced or metastatic malignancy with an NTRK1, NTRK2, or NTRK3 gene amplification identified through molecular assays (such as IHC and any next-generation sequencing [NGS] platform, reference lab NGS, or in house NGS platform) as routinely performed at The University of Texas MD Anderson Cancer Center or other similarly-certified laboratories. The minimum level of amplification is 7 copies. This rationale of amplification level is based on data from MOCLIA at The University of Texas MD Anderson Cancer Center
* Must have received prior standard therapy appropriate for tumor type and stage of disease, or, in the opinion of the investigator, is unlikely to tolerate or derive clinically meaningful benefit from appropriate standard of care therapy
* Must have at least one measurable lesion as defined by RECIST v1.1. Subjects with primary CNS tumors should meet the following criteria:

  * Must have received prior treatment including radiation and/or chemotherapy, with radiation completed > 12 weeks prior to cycle 1 day 1 (C1D1) of therapy, as recommended or appropriate for the tumor type
  * Must have >= 1 site of bi-dimensionally measurable disease (confirmed by magnetic resonance imaging [MRI] and evaluable by RANO), with the size of at least one of the measurable lesions >= 1 cm in each dimension
  * Must have imaging study within 28 days before enrollment. If on steroid therapy, the dose must be stable for at least five days immediately before and during the imaging study
* Eastern Cooperative Oncology Group (ECOG) score =< 3. If enrolled with primary CNS tumor to be assessed by RANO, Karnofsky performance score (KPS) >= 70 %
* Archived tumor tissue. If archival tissue is unavailable, an on-study tumor biopsy should be attempted if it can be safely performed
* Serum aspartate aminotransferase (AST) and serum alanine aminotransferase (ALT) < 2.5 x upper limit of normal (ULN) or < 5 x ULN if liver function abnormalities are due to underlying malignancy
* Total bilirubin < 2.5 x ULN, except in cases of biliary obstruction. Subjects with a known history of Gilberts disease and an isolated elevation of indirect bilirubin are eligible
* Serum creatinine < 2.0 x ULN or estimated glomerular filtration rate >= 30 mL/minute using the Cockcroft-Gault formula
* Ability to comply with outpatient treatment, laboratory monitoring, and required clinic visits for the duration of study participation
* Willingness of men and women of reproductive potential to use two effective birth control methods, one used by the subject and another by his/her partner, for the duration of treatment and for 3 months following study completion

Exclusion Criteria:

* Investigational agent or anticancer therapy within 2 weeks prior to the planned start of larotrectinib or five half-lives, whichever is shorter, and without clinically significant toxicities from that therapy
* Prior progression while receiving approved or investigational tyrosine kinase inhibitors targeting TRK. However, subjects who received less than 28 days of such treatment and discontinued because of intolerance or toxicity are eligible
* Symptomatic or unstable brain metastases that needs corticosteroid usage. Subjects with asymptomatic brain metastases or primary CNS tumors are eligible
* Uncontrolled concurrent malignancy that would limit assessment of efficacy. Allowed diseases may include, but are not limited to in situ cancers of cervix, breast, or skin, superficial bladder cancer, limited-stage prostate cancer, and basal or squamous cancers of the skin
* Active uncontrolled systemic bacterial, viral, or fungal infection, unstable cardiovascular disease or other systemic disease that would limit compliance with study procedures. Unstable cardiovascular disease is defined as:

  * Persistently uncontrolled hypertension defined as systolic blood pressure (BP) > 150 mmHg and/or diastolic BP > 100 mmHg despite antihypertensive therapy
  * Myocardial infarction within 3 months of screening
* Stroke within 3 months of screening
* Inability to discontinue treatment with a strong cytochrome P450 (CYP450), 3A4 (CYP3A4) inhibitor or inducer prior to start of treatment
* Pregnancy or lactation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2027-11-11 (Estimated); Study Completion 2027-11-11 (Estimated)

PRIMARY OUTCOMES:
Overall response | Up to 2 years post-treatment
  Will be scored by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Best overall response of confirmed complete response or partial response | Up to 2 years post-treatment
  Will be determined using RECIST version 1.1 or Response Assessment in Neuro-Oncology criteria, as appropriate to tumor type. A bias-correcting estimate of the best overall response rate and its one-sided 90% confidence interval will be calculated using an exact inference method that appropriately accounts for Bayesian optimal phase II design.
Duration of response | From the date complete response or partial response is first noted (whichever response is recorded first), to the date that recurrence or progressive disease is first documented or to date of death, assessed up to 2 years
  Will be calculated for subjects who achieve confirmed complete response or partial response, and Kaplan-Meier estimates, mean and median duration, and two-sided 95% confidence intervals will be generated.
Growth modulation index | Up to 2 years post-treatment
  Will be defined as the ratio of time to progression (TTP) with nth line of therapy (TTPn) to the most recent prior line of therapy and summarized with mean, median, standard error, and two-sided 95% confidence interval.
Progression-free survival | From initiation of larotrectinib to disease progression or death due to any cause, whichever occurs first, assessed up to 2 years
  Kaplan-Meier estimates, mean and median duration, and two-sided 95% confidence intervals will be generated. In patients who have received prior therapy, corresponding Kaplan-Meier plots, mean and median duration with 95% confidence intervals will be used to compare the duration of progression-free survival following initiation of larotrectinib to that following the line of therapy immediately preceding larotrectinib.
Overall survival | From initiation of treatment to death from any cause, assessed up to 2 years
  Kaplan-Meier estimates, mean and median duration, and two-sided 95% confidence intervals will be generated.
Clinical benefit rate | Up to 2 years post-treatment
  Will be defined as the proportion of subjects with best overall response of complete response, partial response, or stable disease lasting 16 or more weeks following initiation of treatment and summarized in percentages with two-sided 95% confidence intervals.
Incidence of adverse events | Up to 4 weeks (after the final dose of the last cycle of treatment (between 21 and 35 days)
  Safety will be assessed by clinical review of all relevant parameters including adverse events, serious adverse events, laboratory values, vital signs, and electrocardiogram results. Overall safety profiles will be provided along with tumor-specific profiles. Treatment-emergent adverse events, defined as adverse events that start on or after the first administration of study drug, will be summarized based on the number and percentage of subjects experiencing the event, as defined by Medical Dictionary for Regulatory Activities system organ class and preferred term. In the event a subject experiences repeat episodes of the same adverse event, then the event with the highest severity grade and strongest causal relationship to study drug will be used for purposes of incidence tabulations.
Change in clinical safety laboratory values and vital signs | Baseline up to 2 years post-treatment
  Waterfall plots will be used to depict graphically for individual subjects the maximum percentage decrease from baseline in the sum of the longest diameters of target lesions. Similarly, spider and swimmer plots will be used to display the change in tumor burden over time for individual subjects and the occurrence of clinical outcomes of interest (e.g., tumor response, disease progression, treatment discontinuation, death).

CONTACTS AND LOCATIONS:
Overall Officials: David S Hong, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States